CLINICAL TRIAL: NCT01519089
Title: A Phase 3, Multi Site, Randomized, Double Blind Study Of The Long-term Safety, Tolerability And Efficacy Of 2 Oral Doses Of Cp 690,550 In Subjects With Moderate To Severe Plaque Psoriasis And/or Psoriatic Arthritis
Brief Title: A Long Term Study To Evaluate The Safety, Tolerability And Efficacy Of CP-690,550 In Patients With Moderate To Severe Plaque Psoriasis And/Or Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921137
Record Dates: First submitted 2011-12-22; First posted 2012-01-26 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Psoriasis
Keywords: chronic; severe; moderate; treatment; safety; efficacy; CP-690; 550; Plaque psoriasis; Psoriasis Vulgaris; Psoriatic Arthritis; tofacitinib; Xeljanz
MeSH Terms: conditions — Psoriasis; Bronchiolitis Obliterans Syndrome; Lymphoma, Follicular; Arthritis, Psoriatic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CP-690,550 10 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- CP690,550 5 mg BID (Experimental)
  Interventions: Drug: CP-690, 550

INTERVENTIONS:
Drug: CP-690,550 — 10 mg BID, continuous treatment for 16 weeks under blinding, 10 mg BID, continuous treatment for 4 weeks and variable dose (5 mg or 10 mg), continuous treatment for 32 weeks.
  Arms: CP-690,550 10 mg BID
Drug: CP-690, 550 — 5 mg BID, continuous treatment for 16 weeks under blinding, 10 mg BID, continuous treatment for 4 weeks and variable dose (5 mg or 10 mg), continuous treatment for 32 weeks.
  Arms: CP690,550 5 mg BID

SUMMARY:
The main objective of this study is to evaluate the long term safety of CP-690,550 in patients being treated for moderate to severe plaque psoriasis and/or psoriatic arthritis. This study will also to compare the efficacy of two oral doses of CP-690,550 (5 mg BID and 10 mg BID) after 16 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Are 20 years or older and considered to be candidates for systemic or phototherapy.

[Moderate to Severe Plaque Psoriasis]

* Diagnosed for at least 12 months.
* Have Psoriasis Area and Severity Index (PASI) score of 12 and plaque type psoriasis covering at least 10% of body surface area (BSA).

[Psoriatic Arthritis]

* Diagnosed for at least 6 months.
* Meet the CASPAR (classification criteria for Psoriatic Arthritis) criteria at screening;
* Have active arthritis (≥3 tender/painful joints on motion and ≥3 swollen joints), and active plaque psoriasis with at least 2 cm in diameter.

Exclusion Criteria:

* Non-plaque or drug induced forms of psoriasis
* Cannot discontinue current oral, injectable or topical therapy for psoriasis/psoriatic arthritis or cannot discontinue phototherapy (PUVA or UVB)
* any uncontrolled significant medical condition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Japan (16):
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - JR Sapporo hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Chuo-ku, Kobe, Hyōgo
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Nissay Hospital, Osaka, Osaka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Teishin Hospital, Chiyoda-ku, Tokyo
  - Tokyo medical university Hachioji medical center, Hachiōji, Tokyo
  - Kanto Medical Center NTT East Corporation, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjyuku-ku, Tokyo
  - Tonami General Hospital, Tonami, Toyama
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Jikei University Hospital, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921137&StudyName=A%20Long%20Term%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%20And%20Efficacy%20Of%20CP-690%2C550%20In%20Patients%20With%20Moderate%20To%20Severe%20Plaque%20Psori

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg BID: CP-690,550 5 mg tablet orally twice daily (BID) up to Week 16: CP-690,550 10 mg BID from Week 16 to 20: variable 5 or 10 mg BID from Week 20 to Week 52.
- CP-690,550 10 mg BID: CP-690,550 10 mg tablet orally twice daily (BID) up to Week 16: CP-690,550 10 mg BID from Week 16 to 20: variable 5 or 10 mg BID from Week 20 to Week 52.
Period: Overall Study
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID
Started | 47 | 48
Received Treatment | 47 | 47
Completed | 40 | 33
Not Completed | 7 | 15
Not completed — Adverse Event | 4 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 2 | 6
Not completed — Not received study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.8) | 46.4 (10.8) | 48.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI75) Response at Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring assessed by the investigator, of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least a 75 percent (%) reduction in PASI at Week 16 relative to Baseline.
Time Frame: Week 16
Population: Moderate to Severe Plaque Psoriasis Population: Participants who met the inclusion criteria for the moderate to severe plaque psoriasis in the Full Analysis Set (FAS). FAS included all participants randomized and treated with at least 1 dose of study drugs. Missing data was imputed as non-responder.
Measure: Number; unit: Percentage of participants
Groups:
- Total: (=sum across Arm/Groups)
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants | 62.8 | 72.7 | 67.8

2. Primary Outcome: Percentage of Participants With a Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear' at Week 16
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear).
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants | 67.4 | 68.2 | 67.8

3. Primary Outcome: Proportion of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 16
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 16
Population: Psoriatic Arthritis Population: Participants who met the inclusion criteria for the psoriatic arthritis in the Full Analysis Set (FAS). FAS included all participants randomized and treated with at least 1 dose of study drugs. Missing data was imputed as non-responder.
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Percentage of participants | 100 | 100 | 100

4. Primary Outcome: Number of Participants With Adjudicated Cardiovacular Events
Description: Adjudicated cardiovascular events were assessed by investigators as independent reviewers based on event documentation including: hospital discharge summaries, operative reports, clinic notes, ECGs, diagnostic enzymes, results of other diagnostic tests, autopsy reports and death certificate information; specific requirements vary with the event requiring adjudication.
Time Frame: Baseline to Follow-up
Population: Participants treated with at least 1 dose of study drugs.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 47 | 47 | 94
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Malignancy Events _Week 0 Through Follow-up
Description: For all biopsies of potentially malignant tumors, suspicious lymphadenopathy, or possible extranodal LPD, the study site requested the pathologist to send the original slides used to make the definitive diagnosis, ancillary study reports, and the pathologist's report to the central laboratory for a blinded review by a central pathologist.
Time Frame: Baseline to Follow-up
Population: Participants treated with at least 1 dose of study drugs.
Measure: Number; unit: Participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 47 | 47 | 94
Participants
  Number of participants with any malignancy events | 0 | 0 | 0
  Malignancy excluding non-melanoma skin cancer | 0 | 0 | 0
  Lymphoma/Lymphoproliferative disorders (LPD) | 0 | 0 | 0
  Melanoma | 0 | 0 | 0
  Non-melanoma skin cancer | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI75) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring assessed by the investigator, of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least a 75 percent (%) reduction in PASI at the each visit relative to Baseline.
Time Frame: Week 2, 4, 8, 12, 20, 28, 40, 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants
  Week 2 | 2.3 | 4.5 | 3.4
  Week 4 | 7.0 | 22.7 | 14.9
  Week 8 | 41.9 | 54.5 | 48.3
  Week 12 | 60.5 | 70.5 | 65.5
  Week 20 | 67.4 | 63.6 | 65.5
  Week 28 | 69.8 | 65.9 | 67.8
  Week 40 | 69.8 | 63.6 | 66.7
  Week 52 | 62.8 | 63.6 | 63.2

7. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 50 (PASI50) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring assessed by the investigator, of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI50 response was defined as at least a 50 percent (%) reduction in PASI at the each visit relative to Baseline.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants
  Week 2 | 9.3 | 22.7 | 16.1
  Week 4 | 34.9 | 56.8 | 46.0
  Week 8 | 60.5 | 81.8 | 71.3
  Week 12 | 81.4 | 84.1 | 82.8
  Week 16 | 76.7 | 79.5 | 78.2
  Week 20 | 79.1 | 75.0 | 77.0
  Week 28 | 90.7 | 72.7 | 81.6
  Week 40 | 88.4 | 79.5 | 83.9
  Week 52 | 90.7 | 68.2 | 79.3

8. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI90) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring assessed by the investigator, of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI90 response was defined as at least a 90 percent (%) reduction in PASI at the each visit relative to Baseline.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants
  Week 2 | 0.0 | 0.0 | 0.0
  Week 4 | 4.7 | 13.6 | 9.2
  Week 8 | 16.3 | 29.5 | 23.0
  Week 12 | 37.2 | 45.5 | 41.4
  Week 16 | 37.2 | 54.5 | 46.0
  Week 20 | 58.1 | 56.8 | 57.5
  Week 28 | 55.8 | 45.5 | 50.6
  Week 40 | 58.1 | 47.7 | 52.9
  Week 52 | 51.2 | 47.7 | 49.4

9. Secondary Outcome: Time to Achieve a Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear'
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). Median time to achieve a PGA response up to week 16 is reported. The median time to event is estimated based on Kaplan-Meier product-limit method. Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Week 16
Population: Moderate to Severe Plaque Psoriasis Population: Participants who met the inclusion criteria for the moderate to severe plaque psoriasis in the Full Analysis Set (FAS). FAS included all participants randomized and treated with at least 1 dose of study drugs.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Week | 8.0 [8.0 to 12.0] | 8.0 [4.0 to 12.0] | 8.0 [NA to NA] — The 95 percent confidence interval could not be constructed.

10. Secondary Outcome: Time to Achieve a Psoriasis Area and Severity Index 75 (PASI75) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least 75% reduction in PASI relative to Baseline. The median time to event is estimated based on Kaplan-Meier product-limit method. Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Week 16
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Week | 12.0 [8.0 to 16.0] | 8.0 [8.0 to 12.0] | 12.0 [8.0 to 12.0]

11. Secondary Outcome: Time to Achieve a Psoriasis Area and Severity Index 50 (PASI50) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring assessed by the investigator, of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI50 response was defined as at least 50% reduction in PASI relative to Baseline. The median time to event is estimated based on Kaplan-Meier product-limit method. Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Week 16
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Week | 8.0 [4.0 to 12.0] | 4.0 [4.0 to 8.0] | 8.0 [4.0 to 8.0]

12. Secondary Outcome: Time to Achieve a Psoriasis Area and Severity Index 90 (PASI90) Response
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and "percent of BSA" affected. PASI is a composite scoring assessed by the investigator, of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI90 response was defined as at least 90% reduction in PASI relative to Baseline. The median time to event is estimated based on Kaplan-Meier product-limit method. Median time to event is not estimable if the estimated probability of response by Week 16 is less than 50%.
Time Frame: Week 16
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Week | NA [12.0 to NA] — The median time could not be computed because fewer than half of the subjects achieved a PASI90 response. | 12.0 [12.0 to 16.0] | 16.0 [12.0 to NA] — The 95 percent upper limit could not be computed due to the limited analysis duration up to Week 16.

13. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index (PASI) Score >= 125 Percent of the Baseline PASI Score
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants
  Week 2 | 2.3 | 0.0 | 1.1
  Week 4 | 0.0 | 2.3 | 1.1
  Week 8 (n=43, 41, 84) | 0.0 | 0.0 | 0.0
  Week 12 (n=43, 41, 84) | 0.0 | 2.4 | 1.2
  Week 16 (n=43, 40, 83) | 0.0 | 2.5 | 1.2
  Week 20 (n=43, 39, 82) | 0.0 | 0.0 | 0.0
  Week 28 (n=43, 39, 82) | 0.0 | 0.0 | 0.0
  Week 40 (n=41, 38, 79) | 0.0 | 0.0 | 0.0
  Week 52 (n=39, 32, 71) | 0.0 | 0.0 | 0.0

14. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: as for outcome 13
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Units on a scale
  Week 2 | -5.18 (5.898) | -7.36 (6.428) | -6.28 (6.232)
  Week 4 | -10.40 (7.518) | -13.16 (8.739) | -11.79 (8.229)
  Week 8 (n=43, 41, 84) | -15.95 (8.392) | -19.90 (10.741) | -17.88 (9.756)
  Week 12 (n=43, 41, 84) | -18.91 (8.918) | -21.68 (11.598) | -20.26 (10.344)
  Week 16 (n=43, 40, 83) | -19.53 (9.094) | -22.06 (12.606) | -20.75 (10.935)
  Week 20 (n=43, 39, 82) | -20.95 (9.239) | -22.18 (12.045) | -21.53 (10.617)
  Week 28 (n=43, 39, 82) | -21.77 (10.196) | -21.46 (10.503) | -21.62 (10.280)
  Week 40 (n=41, 38, 79) | -22.20 (10.181) | -21.18 (10.229) | -21.71 (10.151)
  Week 52 (n=39, 32, 71) | -21.96 (9.621) | -22.11 (10.598) | -22.03 (10.000)

15. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Component Score
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. Basic characteristics of psoriatic lesions: erythema, induration, and scaling (PASI components) are scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]) according to a 5-point scale: 0 (no involvement); 1 (slight); 2 (moderate); 3 (marked); 4 (very marked). PASI component score range from 0 to 4, where higher scores indicate greater severity of psoriatic lesions.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Units on a scale
  Week 2: Erythema (Head/Neck) | -0.5 (0.83) | -0.9 (0.82) | -0.7 (0.84)
  Week 2: Erythema (Upper Limbs) | -0.5 (0.67) | -0.8 (0.72) | -0.6 (0.70)
  Week 2: Erythema (Trunk) | -0.6 (0.67) | -0.8 (0.69) | -0.7 (0.69)
  Week 2: Erythema (Lower Limbs) | -0.7 (0.69) | -0.8 (0.71) | -0.7 (0.70)
  Week 2: Induration (Head/Neck) | -0.4 (0.70) | -0.8 (0.89) | -0.6 (0.82)
  Week 2: Induration (Upper Limbs) | -0.5 (0.63) | -0.6 (0.75) | -0.6 (0.69)
  Week 2: Induration (Trunk) | -0.5 (0.63) | -0.7 (0.59) | -0.6 (0.62)
  Week 2: Induration (Lower Limbs) | -0.5 (0.67) | -0.7 (0.71) | -0.6 (0.69)
  Week 2: Scaling (Head/Neck) | -0.4 (0.66) | -0.9 (0.91) | -0.7 (0.83)
  Week 2: Scaling (Upper Limbs) | -0.4 (0.59) | -0.8 (0.74) | -0.6 (0.69)
  Week 2: Scaling (Trunk) | -0.3 (0.57) | -0.8 (0.76) | -0.6 (0.71)
  Week 2: Scaling (Lower Limbs) | -0.4 (0.70) | -0.7 (0.73) | -0.6 (0.73)
  Week 4: Erythema (Head/Neck) | -0.8 (1.02) | -1.3 (0.99) | -1.0 (1.02)
  Week 4: Erythema (Upper Limbs) | -1.1 (0.81) | -1.2 (0.94) | -1.1 (0.87)
  Week 4: Erythema (Trunk) | -1.0 (0.64) | -1.3 (0.79) | -1.1 (0.72)
  Week 4: Erythema (Lower Limbs) | -1.1 (0.91) | -1.2 (0.79) | -1.2 (0.85)
  Week 4: Induration (Head/Neck) | -0.7 (0.89) | -1.2 (1.09) | -1.0 (1.02)
  Week 4: Induration (Upper Limbs) | -1.1 (0.86) | -1.0 (0.85) | -1.0 (0.85)
  Week 4: Induration (Trunk) | -0.9 (0.80) | -1.3 (0.82) | -1.1 (0.83)
  Week 4: Induration (Lower Limbs) | -1.0 (0.90) | -1.2 (0.98) | -1.1 (0.94)
  Week 4: Scaling (Head/Neck) | -0.8 (0.86) | -1.2 (0.99) | -1.0 (0.95)
  Week 4: Scaling (Upper Limbs) | -0.9 (0.70) | -1.2 (0.86) | -1.0 (0.79)
  Week 4: Scaling (Trunk) | -0.9 (0.71) | -1.3 (0.95) | -1.1 (0.87)
  Week 4: Scaling (Lower Limbs) | -0.8 (0.72) | -1.3 (0.96) | -1.1 (0.89)
  Week 8: Erythema (Head/Neck) (n=43, 41, 84) | -1.4 (1.13) | -1.6 (1.03) | -1.5 (1.08)
  Week 8: Erythema (Upper Limbs) (n=43, 41, 84) | -1.5 (0.93) | -1.6 (0.98) | -1.5 (0.95)
  Week 8: Erythema (Trunk) (n=43, 41, 84) | -1.7 (0.91) | -1.9 (0.93) | -1.8 (0.92)
  Week 8: Erythema (Lower Limbs) (n=43, 41, 84) | -1.5 (0.91) | -1.7 (0.91) | -1.6 (0.91)
  Week 8: Induration (Head/Neck) (n=43, 41, 84) | -1.3 (0.91) | -1.6 (1.10) | -1.4 (1.01)
  Week 8: Induration (Upper Limbs) (n=43, 41, 84) | -1.6 (0.93) | -1.6 (0.89) | -1.6 (0.91)
  Week 8: Induration (Trunk) (n=43, 41, 84) | -1.6 (0.98) | -1.7 (1.03) | -1.7 (1.00)
  Week 8: Induration (Lower Limbs) (n=43, 41, 84) | -1.6 (0.91) | -1.7 (0.98) | -1.7 (0.94)
  Week 8: Scaling (Head/Neck) (n=43, 41, 84) | -1.3 (0.90) | -1.5 (1.03) | -1.4 (0.96)
  Week 8: Scaling (Upper Limbs) (n=43, 41, 84) | -1.3 (0.80) | -1.6 (0.86) | -1.5 (0.84)
  Week 8: Scaling (Trunk) (n=43, 41, 84) | -1.4 (0.82) | -1.8 (1.00) | -1.6 (0.93)
  Week 8: Scaling (Lower Limbs) (n=43, 41, 84) | -1.3 (0.82) | -1.8 (0.88) | -1.5 (0.88)
  Week 12: Erythema (Head/Neck) (n=43, 41, 84) | -1.7 (1.10) | -1.7 (0.98) | -1.7 (1.04)
  Week 12: Erythema (Upper Limbs) (n=43, 41, 84) | -1.9 (0.99) | -1.8 (1.13) | -1.8 (1.05)
  Week 12: Erythema (Trunk) (n=43, 41, 84) | -2.1 (1.08) | -2.0 (0.95) | -2.0 (1.01)
  Week 12: Erythema (Lower Limbs) (n=43, 41, 84) | -1.9 (0.92) | -1.9 (0.94) | -1.9 (0.92)
  Week 12: Induration (Head/Neck) (n=43, 41, 84) | -1.5 (0.94) | -1.6 (1.12) | -1.6 (1.02)
  Week 12: Induration (Upper Limbs) (n=43, 41, 84) | -1.7 (0.94) | -1.8 (0.99) | -1.7 (0.96)
  Week 12: Induration (Trunk) (n=43, 41, 84) | -2.0 (1.01) | -2.0 (1.00) | -2.0 (1.00)
  Week 12: Induration (Lower Limbs) (n=43, 41, 84) | -1.9 (0.91) | -1.9 (1.06) | -1.9 (0.98)
  Week 12: Scaling (Head/Neck) (n=43, 41, 84) | -1.7 (0.92) | -1.6 (1.02) | -1.6 (0.96)
  Week 12: Scaling (Upper Limbs) (n=43, 41, 84) | -1.4 (0.91) | -1.7 (0.95) | -1.6 (0.94)
  Week 12: Scaling (Trunk) (n=43, 41, 84) | -1.6 (1.05) | -1.9 (1.00) | -1.7 (1.03)
  Week 12: Scaling (Lower Limbs) (n=43, 41, 84) | -1.5 (0.85) | -1.9 (1.00) | -1.7 (0.95)
  Week 16: Erythema (Head/Neck) (n=43, 40, 83) | -1.7 (1.14) | -1.7 (1.07) | -1.7 (1.10)
  Week 16: Erythema (Upper Limbs) (n=43, 40, 83) | -1.9 (1.13) | -1.9 (1.12) | -1.9 (1.12)
  Week 16: Erythema (Trunk) (n=43, 40, 83) | -2.1 (1.10) | -2.0 (1.07) | -2.0 (1.08)
  Week 16: Erythema (Lower Limbs) (n=43, 40, 83) | -2.0 (1.03) | -1.9 (0.94) | -2.0 (0.99)
  Week 16: Induration (Head/Neck) (n=43, 40, 83) | -1.5 (0.96) | -1.6 (1.17) | -1.6 (1.06)
  Week 16: Induration (Upper Limbs) (n=43, 40, 83) | -1.8 (0.96) | -1.8 (1.01) | -1.8 (0.98)
  Week 16: Induration (Trunk) (n=43, 40, 83) | -2.1 (1.01) | -2.0 (1.01) | -2.0 (1.01)
  Week 16: Induration (Lower Limbs) (n=43, 40, 83) | -2.1 (0.95) | -2.0 (1.08) | -2.0 (1.01)
  Week 16: Scaling (Head/Neck) (n=43, 40, 83) | -1.6 (0.95) | -1.6 (1.08) | -1.6 (1.01)
  Week 16: Scaling (Upper Limbs) (n=43, 40, 83) | -1.5 (0.93) | -1.7 (1.05) | -1.6 (0.99)
  Week 16: Scaling (Trunk) (n=43, 40, 83) | -1.6 (0.96) | -1.8 (1.09) | -1.7 (1.02)
  Week 16: Scaling (Lower Limbs) (n=43, 40, 83) | -1.6 (0.93) | -1.8 (1.06) | -1.7 (1.00)
  Week 20: Erythema (Head/Neck) (n=43, 39, 82) | -1.8 (1.15) | -1.6 (0.96) | -1.7 (1.07)
  Week 20: Erythema (Upper Limbs) (n=43, 39, 82) | -1.9 (0.97) | -1.9 (1.26) | -1.9 (1.11)
  Week 20: Erythema (Trunk) (n=43, 39, 82) | -2.2 (1.04) | -2.1 (1.04) | -2.1 (1.04)
  Week 20: Erythema (Lower Limbs) (n=43, 39, 82) | -2.1 (1.04) | -2.1 (1.09) | -2.1 (1.05)
  Week 20: Induration (Head/Neck) (n=43, 39, 82) | -1.6 (1.00) | -1.5 (1.12) | -1.6 (1.06)
  Week 20: Induration (Upper Limbs) (n=43, 39, 82) | -1.9 (0.97) | -1.7 (1.14) | -1.8 (1.05)
  Week 20: Induration (Trunk) (n=43, 39, 82) | -2.1 (1.01) | -1.9 (1.07) | -2.0 (1.04)
  Week 20: Induration (Lower Limbs) (n=43, 39, 82) | -2.2 (0.95) | -2.0 (1.06) | -2.1 (1.00)
  Week 20: Scaling (Head/Neck) (n=43, 39, 82) | -1.7 (0.94) | -1.5 (1.05) | -1.6 (0.99)
  Week 20: Scaling (Upper Limbs) (n=43, 39, 82) | -1.5 (0.96) | -1.6 (1.14) | -1.5 (1.04)
  Week 20: Scaling (Trunk) (n=43, 39, 82) | -1.7 (0.93) | -1.8 (1.05) | -1.8 (0.99)
  Week 20: Scaling (Lower Limbs) (n=43, 39, 82) | -1.7 (0.92) | -1.8 (1.16) | -1.8 (1.04)
  Week 28: Erythema (Head/Neck) (n=43, 39, 82) | -1.8 (1.11) | -1.6 (0.81) | -1.7 (0.98)
  Week 28: Erythema (Upper Limbs) (n=43, 39, 82) | -2.1 (1.09) | -1.8 (1.07) | -2.0 (1.08)
  Week 28: Erythema (Trunk) (n=43, 39, 82) | -2.1 (1.13) | -2.0 (0.99) | -2.1 (1.06)
  Week 28: Erythema (Lower Limbs) (n=43, 39, 82) | -2.3 (1.05) | -1.9 (0.99) | -2.1 (1.03)
  Week 28: Induration (Head/Neck) (n=43, 39, 82) | -1.7 (0.97) | -1.6 (0.99) | -1.6 (0.98)
  Week 28: Induration (Upper Limbs) (n=43, 39, 82) | -2.0 (1.12) | -1.7 (1.10) | -1.9 (1.12)
  Week 28: Induration (Trunk) (n=43, 39, 82) | -2.0 (1.12) | -1.8 (1.16) | -1.9 (1.14)
  Week 28: Induration (Lower Limbs) (n=43, 39, 82) | -2.2 (1.03) | -1.8 (1.14) | -2.0 (1.09)
  Week 28: Scaling (Head/Neck) (n=43, 39, 82) | -1.7 (1.01) | -1.4 (1.07) | -1.6 (1.04)
  Week 28: Scaling (Upper Limbs) (n=43, 39, 82) | -1.8 (1.05) | -1.6 (1.02) | -1.7 (1.03)
  Week 28: Scaling (Trunk) (n=43, 39, 82) | -1.7 (0.99) | -1.8 (1.11) | -1.7 (1.05)
  Week 28: Scaling (Lower Limbs) (n=43, 39, 82) | -1.8 (1.09) | -1.7 (1.02) | -1.7 (1.05)
  Week 40: Erythema (Head/Neck) (n=41, 38, 79) | -1.9 (1.10) | -1.7 (0.90) | -1.8 (1.01)
  Week 40: Erythema (Upper Limbs) (n=41, 38, 79) | -2.1 (1.05) | -1.9 (1.06) | -2.0 (1.06)
  Week 40: Erythema (Trunk) (n=41, 38, 79) | -2.1 (1.04) | -2.2 (0.87) | -2.2 (0.95)
  Week 40: Erythema (Lower Limbs) (n=41, 38, 79) | -2.4 (1.05) | -2.0 (1.03) | -2.2 (1.05)
  Week 40: Induration (Head/Neck) (n=41, 38, 79) | -1.7 (1.05) | -1.5 (1.08) | -1.6 (1.07)
  Week 40: Induration (Upper Limbs) (n=41, 38, 79) | -2.0 (1.18) | -1.8 (0.98) | -1.9 (1.09)
  Week 40: Induration (Trunk) (n=41, 38, 79) | -1.9 (1.26) | -2.1 (0.93) | -2.1 (1.11)
  Week 40: Induration (Lower Limbs) (n=41, 38, 79) | -2.2 (1.14) | -1.9 (1.03) | -2.1 (1.10)
  Week 40: Scaling (Head/Neck) (n=41, 38, 79) | -1.8 (0.97) | -1.4 (1.00) | -1.6 (0.99)
  Week 40: Scaling (Upper Limbs) (n=41, 38, 79) | -1.7 (1.10) | -1.8 (0.94) | -1.7 (1.02)
  Week 40: Scaling (Trunk) (n=41, 38, 79) | -1.7 (0.93) | -1.9 (1.03) | -1.8 (0.98)
  Week 40: Scaling (Lower Limbs) (n=41, 38, 79) | -1.9 (1.11) | -1.8 (1.06) | -1.8 (1.08)
  Week 52: Erythema (Head/Neck) (n=39, 32, 71) | -1.9 (1.17) | -1.6 (1.24) | -1.8 (1.20)
  Week 52: Erythema (Upper Limbs) (n=39, 32, 71) | -2.0 (1.15) | -2.0 (0.90) | -2.0 (1.04)
  Week 52: Erythema (Trunk) (n=39, 32, 71) | -2.2 (1.01) | -2.2 (0.93) | -2.2 (0.97)
  Week 52: Erythema (Lower Limbs) (n=39, 32, 71) | -2.1 (1.11) | -2.2 (0.94) | -2.1 (1.03)
  Week 52: Induration (Head/Neck) (n=39, 32, 71) | -1.7 (1.06) | -1.5 (1.22) | -1.6 (1.13)
  Week 52: Induration (Upper Limbs) (n=39, 32, 71) | -1.9 (1.21) | -2.0 (0.97) | -1.9 (1.10)
  Week 52: Induration (Trunk) (n=39, 32, 71) | -1.8 (1.39) | -2.1 (1.03) | -2.0 (1.24)
  Week 52: Induration (Lower Limbs) (n=39, 32, 71) | -2.0 (1.29) | -2.2 (0.97) | -2.1 (1.15)
  Week 52: Scaling (Head/Neck) (n=39, 32, 71) | -1.8 (0.98) | -1.6 (1.08) | -1.7 (1.02)
  Week 52: Scaling (Upper Limbs) (n=39, 32, 71) | -1.6 (1.02) | -1.9 (0.98) | -1.7 (1.01)
  Week 52: Scaling (Trunk) (n=39, 32, 71) | -1.6 (0.96) | -1.9 (1.01) | -1.7 (0.98)
  Week 52: Scaling (Lower Limbs) (n=39, 32, 71) | -1.7 (1.15) | -2.0 (1.03) | -1.8 (1.10)

16. Secondary Outcome: Percentage of Participants With a Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear'
Description: as for outcome 2
Time Frame: Week 2, 4, 8, 12, 20, 28, 40, 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants
  Week 2 | 7.0 | 15.9 | 11.5
  Week 4 | 30.2 | 38.6 | 34.5
  Week 8 | 58.1 | 61.4 | 59.8
  Week 12 | 72.1 | 75.0 | 73.6
  Week 20 | 72.1 | 59.1 | 65.5
  Week 28 | 67.4 | 54.5 | 60.9
  Week 40 | 67.4 | 54.5 | 60.9
  Week 52 | 58.1 | 56.8 | 57.5

17. Secondary Outcome: Percentage of Participants in a Physician Global Assessment (PGA) of Psoriasis Score Category
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe).
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants
  Week 2: Clear | 0 | 0 | 0
  Week 2: Almost Clear | 7.0 | 15.9 | 11.5
  Week 2: Mild | 39.5 | 43.2 | 41.4
  Week 2: Moderate | 46.5 | 34.1 | 40.2
  Week 2: Severe | 7.0 | 6.8 | 6.9
  Week 4: Clear | 0 | 11.4 | 5.7
  Week 4: Almost Clear | 30.2 | 27.3 | 28.7
  Week 4: Mild | 44.2 | 40.9 | 42.5
  Week 4: Moderate | 18.6 | 20.5 | 19.5
  Week 4: Severe | 7.0 | 0 | 3.4
  Week 8: Clear (n=43, 41, 84) | 7.0 | 26.8 | 16.7
  Week 8: Almost Clear (n=43, 41, 84) | 51.2 | 39.0 | 45.2
  Week 8: Mild (n=43, 41, 84) | 27.9 | 24.4 | 26.2
  Week 8: Moderate (n=43, 41, 84) | 14.0 | 9.8 | 11.9
  Week 8: Severe (n=43, 41, 84) | 0 | 0 | 0
  Week 12: Clear (n=43, 41, 84) | 14.0 | 36.6 | 25.0
  Week 12: Almost Clear (n=43, 41, 84) | 58.1 | 43.9 | 51.2
  Week 12: Mild (n=43, 41, 84) | 20.9 | 9.8 | 15.5
  Week 12: Moderate (n=43, 41, 84) | 7.0 | 9.8 | 8.3
  Week 12: Severe (n=43, 41, 84) | 0 | 0 | 0
  Week 16: Clear (n=43, 40, 83) | 27.9 | 40.0 | 33.7
  Week 16: Almost Clear (n=43, 40, 83) | 39.5 | 35.0 | 37.3
  Week 16: Mild (n=43, 40, 83) | 25.6 | 17.5 | 21.7
  Week 16: Moderate (n=43, 40, 83) | 7.0 | 5.0 | 6.0
  Week 16: Severe (n=43, 40, 83) | 0 | 2.5 | 1.2
  Week 20: Clear (n=43, 39, 82) | 27.9 | 38.5 | 32.9
  Week 20: Almost Clear (n=43, 39, 82) | 44.2 | 28.2 | 36.6
  Week 20: Mild (n=43, 39, 82) | 18.6 | 25.6 | 22.0
  Week 20: Moderate (n=43, 39, 82) | 9.3 | 7.7 | 8.5
  Week 20: Severe(n=43, 39, 82) | 0 | 0 | 0
  Week 28: Clear (n=43, 39, 82) | 37.2 | 33.3 | 35.4
  Week 28: Almost Clear (n=43, 39, 82) | 30.2 | 28.2 | 29.3
  Week 28: Mild (n=43, 39, 82) | 27.9 | 30.8 | 29.3
  Week 28: Moderate (n=43, 39, 82) | 4.7 | 7.7 | 6.1
  Week 28: Severe (n=43, 39, 82) | 0 | 0 | 0
  Week 40: Clear (n=41, 38, 79) | 43.9 | 34.2 | 39.2
  Week 40: Almost Clear (n=41, 38, 79) | 26.8 | 28.9 | 27.8
  Week 40: Mild (n=41, 38, 79) | 24.4 | 28.9 | 26.6
  Week 40: Moderate (n=41, 38, 79) | 4.9 | 7.9 | 6.3
  Week 40: Severe (n=41, 38, 79) | 0 | 0 | 0
  Week 52: Clear (n=39, 32, 71) | 41.0 | 43.8 | 42.3
  Week 52: Almost Clear (n=39, 32, 71) | 23.1 | 34.4 | 28.2
  Week 52: Mild (n=39, 32, 71) | 30.8 | 18.8 | 25.4
  Week 52: Moderate (n=39, 32, 71) | 5.1 | 3.1 | 4.2
  Week 52: Severe (n=39, 32, 71) | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants Maintaining Psoriasis Area and Severity Index 75 (PASI75) Response After Week 16
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least a 75 percent (%) reduction in PASI relative to Baseline. Maintenance of PASI75 response at Week 52 among participants achieving PASI75 response at Week 16 is reported.
Time Frame: Week 20, 28, 40, 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 28 | 35 | 63
Percentage of participants
  Week 20 | 96.3 | 87.5 | 91.5
  Week 28 | 92.6 | 78.1 | 84.7
  Week 40 | 81.5 | 71.9 | 76.3
  Week 52 | 70.4 | 62.5 | 66.1

19. Secondary Outcome: Percentage of Participants Maintaining Physician Global Assessment (PGA) of Psoriasis Score of 'Clear' or 'Almost Clear'
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). Maintenance of PGA response at Week 52 among participants achieving PGA response at Week 16 is reported.
Time Frame: Week 20, 28, 40, 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 30 | 31 | 61
Percentage of participants
  Week 20 | 100 | 83.3 | 91.5
  Week 28 | 93.1 | 73.3 | 83.1
  Week 40 | 82.8 | 66.7 | 74.6
  Week 52 | 65.5 | 60.0 | 62.7

20. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores = more severe psoriasis.
Time Frame: Week 8, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 32 | 30 | 62
Units on a scale
  Week 8 (n=32, 28, 60) | -3.3 (9.63) | -1.8 (7.72) | -2.6 (8.75)
  Week 16 (n=32, 28, 60) | -11.2 (15.27) | -9.4 (12.66) | -10.4 (14.02)
  Week 20 (n=32, 27, 59) | -15.0 (15.29) | -14.1 (13.03) | -14.6 (14.18)
  Week 28 (n=32, 27, 59) | -21.1 (15.83) | -16.4 (15.27) | -18.9 (15.62)
  Week 40 (n=31, 26, 57) | -22.2 (16.18) | -16.2 (14.13) | -19.5 (15.45)
  Week 52 (n=30, 22, 52) | -20.6 (15.16) | -16.2 (15.62) | -18.7 (15.36)

21. Secondary Outcome: Number of Affected Nails
Description: Nail psoriasis is evaluated by the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lulunea, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Total number psoriasis affected nails (presence of psoriatic manifestations on the nail matrix/nail bed) were assessed and reported.
Time Frame: Baseline, Week 8, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nails
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 32 | 30 | 62
nails
  Baseline | 7.94 (2.82) | 7.13 (3.07) | 7.55 (2.95)
  Week 8 (n=32, 28, 60) | 7.66 (3.17) | 7.11 (3.02) | 7.40 (3.09)
  Week 16 (n=32, 28, 60) | 6.91 (3.43) | 5.75 (3.56) | 6.37 (3.51)
  Week 20 (n=32, 27, 59) | 6.16 (3.60) | 4.59 (4.02) | 5.44 (3.85)
  Week 28 (n=32, 27, 59) | 4.53 (3.87) | 3.59 (3.96) | 4.10 (3.91)
  Week 40 (n=31, 26, 57) | 3.32 (3.94) | 3.77 (3.81) | 3.53 (3.85)
  Week 52 (n=30, 22, 52) | 3.73 (4.25) | 2.50 (3.07) | 3.21 (3.81)

22. Secondary Outcome: Itch Severity Item (ISI) Score
Description: ISI assessed severity of itch (pruritus) due to psoriasis. ISI is a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends for post baseline time points. Baseline ISI is average of scores on 7 days prior to start of study treatment.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Units on a scale
  Baseline | 6.16 (2.669) | 5.32 (2.967) | 5.74 (2.839)
  Week 2 | 5.19 (2.797) | 3.30 (2.530) | 4.23 (2.815)
  Week 4 | 3.65 (2.379) | 2.27 (2.472) | 2.95 (2.510)
  Week 8 (n=43, 41, 84) | 2.26 (2.381) | 1.22 (1.739) | 1.75 (2.145)
  Week 12 (n=43, 41, 84) | 1.77 (2.379) | 1.20 (1.833) | 1.49 (2.137)
  Week 16 (n=43, 40, 83) | 1.67 (2.378) | 0.90 (1.257) | 1.30 (1.949)
  Week 20 (n=43, 39, 82) | 0.95 (1.618) | 1.28 (1.589) | 1.11 (1.603)
  Week 28 (n=43, 39, 82) | 1.12 (1.651) | 1.62 (2.196) | 1.35 (1.933)
  Week 40 (n=41, 38, 79) | 0.90 (1.814) | 1.13 (1.848) | 1.01 (1.822)
  Week 52 (n=39, 32, 71) | 1.15 (2.084) | 0.91 (1.329) | 1.04 (1.776)

23. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: The DLQI is a 10 item general dermatology questionnaire that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI item response options are rated by the participant from 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Units on a scale
  Baseline | 11.3 (6.25) | 8.6 (5.91) | 9.9 (6.19)
  Week 2 | 7.8 (5.20) | 5.8 (5.32) | 6.8 (5.32)
  Week 4 (n=43, 43, 86) | 5.9 (5.07) | 4.2 (4.63) | 5.1 (4.90)
  Week 8 (n=43, 41, 84) | 4.0 (3.95) | 2.8 (3.30) | 3.4 (3.67)
  Week 12 (n=43, 41, 84) | 2.6 (2.86) | 1.8 (2.68) | 2.2 (2.79)
  Week 16 (n=43, 40, 83) | 2.2 (3.04) | 1.9 (2.73) | 2.1 (2.88)
  Week 20 (n=43, 39, 82) | 1.9 (3.13) | 1.8 (2.54) | 1.9 (2.84)
  Week 28 (n=43, 39, 82) | 1.7 (2.66) | 2.9 (3.68) | 2.3 (3.23)
  Week 40 (n=41, 38, 79) | 1.8 (2.81) | 2.3 (4.11) | 2.0 (3.48)
  Week 52 (n=39, 32, 71) | 1.6 (2.42) | 2.2 (4.00) | 1.9 (3.22)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2, Acute (SF-36): Domain Score
Description: 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects are summarized as physical and mental health summary scores. The score range for the physical and mental health scores is 0-100 (100=highest level of functioning).
Time Frame: Week (W) 16, 28, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Units on a scale
  W16: Physical Functioning Domain (n=43, 40, 83) | 1.951 (5.1880) | 4.809 (9.1822) | 3.329 (7.4800)
  W16: Role-Physical Domain (n=43, 40, 83) | 6.160 (9.3615) | 5.130 (11.1600) | 5.664 (10.2172)
  W16: Bodily Pain Domain (n=43, 40, 83) | 11.808 (13.8431) | 10.663 (12.2936) | 11.256 (13.0524)
  W16: General Health Domain (n=43, 40, 83) | 2.392 (7.0933) | 4.333 (7.0145) | 3.328 (7.0799)
  W16: Vitality Domain (n=43, 40, 83) | 4.664 (9.5406) | 3.517 (11.4421) | 4.112 (10.4509)
  W16: Social Function Domain (n=43, 40, 83) | 7.629 (9.9734) | 7.932 (8.8645) | 7.775 (9.3992)
  W16: Role-Emotional Domain (n=43, 40, 83) | 7.219 (11.5898) | 5.584 (11.5654) | 6.431 (11.5365)
  W16: Mental Health Domain (n=43, 40, 83) | 5.928 (12.8757) | 5.125 (13.3613) | 5.541 (13.0378)
  W28: Physical Functioning Domain (n=43, 39, 82) | 1.571 (6.3446) | 4.303 (10.3695) | 2.870 (8.5558)
  W28: Role-Physical Domain (n=43, 39, 82) | 5.882 (10.6375) | 5.017 (11.4671) | 5.471 (10.9795)
  W28: Bodily Pain Domain (n=43, 39, 82) | 10.113 (15.9485) | 8.394 (12.5405) | 9.295 (14.3670)
  W28: General Health Domain (n=43, 39, 82) | 2.644 (5.9230) | 3.517 (7.1375) | 3.059 (6.5025)
  W28: Vitality Domain (n=43, 39, 82) | 4.038 (10.0116) | 3.608 (10.0742) | 3.833 (9.9815)
  W28: Social Function Domain (n=43, 39, 82) | 6.628 (11.3068) | 6.205 (10.4347) | 6.427 (10.8358)
  W28: Role-Emotional Domain (n=43, 39, 82) | 7.395 (11.8846) | 6.310 (12.9504) | 6.879 (12.3375)
  W28: Mental Health Domain (n=43, 39, 82) | 6.701 (12.4375) | 5.328 (12.8129) | 6.048 (12.5580)
  W52: Physical Functioning Domain (n=39,32,71) | 2.151 (5.6134) | 3.773 (7.3533) | 2.882 (6.4585)
  W52: Role-Physical Domain (n=39, 32, 71) | 6.669 (10.0520) | 4.623 (9.7340) | 5.747 (9.8926)
  W52: Bodily Pain Domain (n=39, 32, 71) | 12.335 (12.1413) | 10.673 (9.7128) | 11.586 (11.0678)
  W52: General Health Domain (n=39, 32, 71) | 2.758 (6.0866) | 4.888 (6.8235) | 3.718 (6.4707)
  W52: Vitality Domain (n=39, 32, 71) | 4.068 (10.5612) | 5.052 (8.5160) | 4.511 (9.6390)
  W52: Social Function Domain (n=39, 32, 71) | 8.411 (9.4598) | 8.402 (9.2577) | 8.407 (9.3024)
  W52: Role-Emotional Domain (n=39, 32, 71) | 8.445 (11.0018) | 5.915 (10.3091) | 7.305 (10.6949)
  W52: Mental Health Domain (n=39, 32, 71) | 7.317 (11.6243) | 6.926 (12.6861) | 7.141 (12.0276)

25. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2, Acute (SF-36): Component Summary Score
Description: as for outcome 24
Time Frame: Week 16, 28, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Units on a scale
  Week 16: Physical Health Score (n=43, 40, 83) | 4.719 (6.6806) | 6.146 (8.5192) | 5.407 (7.6087)
  Week 16: Mental Health Score (n=43, 40, 83) | 6.767 (11.0945) | 5.029 (11.4967) | 5.929 (11.2548)
  Week 28: Physical Health Score (n=43, 39, 82) | 3.770 (7.7829) | 4.799 (8.8893) | 4.259 (8.2914)
  Week 28: Mental Health Score (n=43, 39, 82) | 7.085 (11.3660) | 5.364 (10.9089) | 6.266 (11.1159)
  Week 52: Physical Health Score (n=39, 32, 71) | 4.676 (5.7405) | 5.250 (5.7614) | 4.935 (5.7159)
  Week 52: Mental Health Score (n=39, 32, 71) | 7.878 (10.1983) | 6.826 (10.5988) | 7.404 (10.3192)

26. Secondary Outcome: Work Limitation Questionnaire (WLQ)
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (5 items); Physical Demands scale (6 items); Mental-Interpersonal Demands Scale (9 items); Output Demands Scale (5 items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). The WLQ Index score is the weighted sum of the scores from the 4 WLQ scales (total score: 0 [no loss] to 100 [complete loss of work]).
Time Frame: Baseline (BL), Week (W) 4, 16, 28, 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Units on a scale
  BL: Time Management scale (n=34, 37, 71) | 44.49 (37.783) | 42.36 (33.716) | 43.38 (35.479)
  BL: Physical Demands scale (n=33, 35, 68) | 66.67 (33.522) | 78.40 (31.122) | 72.71 (32.606)
  BL: Mental/Interpersonal Demands Scale(n=34,38,72) | 28.61 (29.012) | 31.52 (30.930) | 30.15 (29.865)
  BL: Output Demands scale (n=33, 37, 70) | 22.61 (26.832) | 30.27 (35.295) | 26.66 (31.602)
  BL: WLQ Index Score (n=34, 38, 72) | 9.55 (6.716) | 10.74 (8.045) | 10.18 (7.420)
  W4: Time Management scale (n=31, 36, 67) | 35.32 (42.425) | 31.39 (36.715) | 33.21 (39.203)
  W4: Physical Demands scale (n=29, 36, 65) | 77.16 (33.013) | 83.59 (29.593) | 80.72 (31.083)
  W4:Mental/Interpersonal Demands Scale(n=32,36,68) | 17.94 (26.979) | 23.39 (32.878) | 20.82 (30.149)
  W4: Output Demands scale (n=30, 36, 66) | 13.50 (21.978) | 20.14 (33.306) | 17.12 (28.704)
  W4: WLQ Index Score (n=32, 37, 69) | 7.23 (5.591) | 8.66 (7.754) | 8.00 (6.827)
  W16: Time Management scale (n=31, 35, 66) | 35.07 (38.894) | 33.29 (39.182) | 34.12 (38.756)
  W16: Physical Demands scale (n=30, 32, 62) | 81.60 (26.982) | 86.52 (25.548) | 84.14 (26.153)
  W16:Mental/Interpersonal Demands Scale(n=31,35,66) | 13.33 (21.038) | 20.28 (33.419) | 17.01 (28.296)
  W16: Output Demands scale (n=32, 33, 65) | 11.88 (20.111) | 19.55 (32.485) | 15.77 (27.175)
  W16: WLQ Index Score (n=32, 35, 67) | 6.88 (4.715) | 8.35 (7.425) | 7.65 (6.276)
  W28: Time Management scale (n=34, 34, 68) | 38.68 (40.100) | 29.78 (39.092) | 34.23 (39.557)
  W28: Physical Demands scale (n=32, 34, 66) | 76.02 (31.041) | 85.42 (24.730) | 80.86 (28.151)
  W28:Mental/Interpersonal Demands Scale(n=33,35,68) | 16.84 (28.242) | 16.39 (27.736) | 16.61 (27.774)
  W28: Output Demands scale (n=33, 34, 67) | 13.94 (27.408) | 14.71 (28.761) | 14.33 (27.892)
  W28: WLQ Index Score (n=34, 36, 70) | 7.43 (6.493) | 7.26 (6.829) | 7.34 (6.620)
  W52: Time Management scale (n=31, 31, 62) | 50.32 (43.683) | 31.88 (40.686) | 41.10 (42.883)
  W52: Physical Demands scale (n=29, 29, 58) | 78.16 (30.205) | 89.74 (24.410) | 83.95 (27.838)
  W52:Mental/Interpersonal Demands Scale(n=30,30,60) | 25.56 (36.007) | 16.89 (27.293) | 21.22 (31.977)
  W52: Output Demands scale (n=30, 29, 59) | 22.63 (33.750) | 12.24 (24.589) | 17.52 (29.813)
  W52: WLQ Index Score (n=32, 31, 63) | 9.44 (8.127) | 7.34 (6.429) | 8.41 (7.358)

27. Secondary Outcome: Percentage of Participants With a Patient Global Assessment (PtGA) of Psoriasis Score Category
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5-point scale (0=clear [no psoriasis]; 1=almost clear; 2=mild; 3=moderate; 4=severe).
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 43 | 44 | 87
Percentage of participants
  Baseline: Clear | 0 | 0 | 0
  Baseline: Almost Clear | 0 | 0 | 0
  Baseline: Mild | 0 | 2.3 | 1.1
  Baseline: Moderate | 41.9 | 43.2 | 42.5
  Baseline: Severe | 58.1 | 54.5 | 56.3
  Week 2: Clear | 0 | 0 | 0
  Week 2: Almost Clear | 2.3 | 0 | 1.1
  Week 2: Mild | 2.3 | 29.5 | 16.1
  Week 2: Moderate | 60.5 | 36.4 | 48.3
  Week 2: Severe | 34.9 | 34.1 | 34.5
  Week 4: Clear (n=43, 43, 86) | 0 | 2.3 | 1.2
  Week 4: Almost Clear (n=43, 43, 86) | 4.7 | 9.3 | 7.0
  Week 4: Mild (n=43, 43, 86) | 18.6 | 25.6 | 22.1
  Week 4: Moderate (n=43, 43, 86) | 53.5 | 48.8 | 51.2
  Week 4: Severe (n=43, 43, 86) | 23.3 | 14.0 | 18.6
  Week 8: Clear (n=43, 41, 84) | 4.7 | 7.3 | 6.0
  Week 8: Almost Clear (n=43, 41, 84) | 14.0 | 17.1 | 15.5
  Week 8: Mild (n=43, 41, 84) | 32.6 | 34.1 | 33.3
  Week 8: Moderate (n=43, 41, 84) | 39.5 | 34.1 | 36.9
  Week 8: Severe (n=43, 41, 84) | 9.3 | 7.3 | 8.3
  Week 12: Clear (n=43, 41, 84) | 2.3 | 7.3 | 4.8
  Week 12: Almost Clear (n=43, 41, 84) | 20.9 | 26.8 | 23.8
  Week 12: Mild (n=43, 41, 84) | 34.9 | 41.5 | 38.1
  Week 12: Moderate (n=43, 41, 84) | 34.9 | 17.1 | 26.2
  Week 12: Severe (n=43, 41, 84) | 7.0 | 7.3 | 7.1
  Week 16: Clear (n=43, 40, 83) | 4.7 | 10.0 | 7.2
  Week 16: Almost Clear (n=43, 40, 83) | 32.6 | 22.5 | 27.7
  Week 16: Mild (n=43, 40, 83) | 23.3 | 35.0 | 28.9
  Week 16: Moderate (n=43, 40, 83) | 32.6 | 22.5 | 27.7
  Week 16: Severe (n=43, 40, 83) | 7.0 | 10.0 | 8.4
  Week 20: Clear (n=43, 39, 82) | 7.0 | 12.8 | 9.8
  Week 20: Almost Clear (n=43, 39, 82) | 37.2 | 23.1 | 30.5
  Week 20: Mild (n=43, 39, 82) | 25.6 | 33.3 | 29.3
  Week 20: Moderate (n=43, 39, 82) | 23.3 | 25.6 | 24.4
  Week 20: Severe (n=43, 39, 82) | 7.0 | 5.1 | 6.1
  Week 28: Clear (n=43, 39, 82) | 11.6 | 5.1 | 8.5
  Week 28: Almost Clear (n=43, 39, 82) | 37.2 | 35.9 | 36.6
  Week 28: Mild (n=43, 39, 82) | 23.3 | 20.5 | 22.0
  Week 28: Moderate (n=43, 39, 82) | 20.9 | 33.3 | 26.8
  Week 28: Severe (n=43, 39, 82) | 7.0 | 5.1 | 6.1
  Week 40: Clear (n=41, 38, 79) | 7.3 | 18.4 | 12.7
  Week 40: Almost Clear (n=41, 38, 79) | 46.3 | 31.6 | 39.2
  Week 40: Mild (n=41, 38, 79) | 19.5 | 18.4 | 19.0
  Week 40: Moderate (n=41, 38, 79) | 22.0 | 26.3 | 24.1
  Week 40: Severe (n=41, 38, 79) | 4.9 | 5.3 | 5.1
  Week 52: Clear (n=39, 32, 71) | 20.5 | 18.8 | 19.7
  Week 52: Almost Clear (n=39, 32, 71) | 20.5 | 31.3 | 25.4
  Week 52: Mild (n=39, 32, 71) | 28.2 | 25.0 | 26.8
  Week 52: Moderate (n=39, 32, 71) | 15.4 | 21.9 | 18.3
  Week 52: Severe (n=39, 32, 71) | 15.4 | 3.1 | 9.9

28. Secondary Outcome: Joint Pain Assessment (JPA)
Description: The JPA assesses severity of joint pain. The JPA is a horizontal numeric rating scale. Participants were asked to "select the number that best describes any joint pain that participant may have experienced over the past 24 hours" with response options ranging from "0-no joint pain" to "10-worst possible joint pain."
Time Frame: Baseline, Week 4, 16, 28, 52
Population: The subjects with a medical history of ongoing psoriatic arthritis (that was defined as the MedDRA preferred term for psoriatic arthropathy regardless of meeting the inclusion criteria for the psoriatic arthritis) in the Full Analysis Set (FAS). FAS included all participants randomized and treated with at least 1 dose of study drugs.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 8 | 15 | 23
Units on a scale
  Baseline | 5.25 (3.327) | 4.60 (2.558) | 4.83 (2.790)
  Week 4 (n=8, 14, 22) | 4.00 (2.726) | 1.36 (1.008) | 2.32 (2.191)
  Week 16 (n=8, 15, 23) | 1.88 (2.295) | 0.60 (0.737) | 1.04 (1.551)
  Week 28 (n=8, 14, 22) | 1.75 (1.753) | 0.86 (0.949) | 1.18 (1.332)
  Week 52 (n=4, 13, 17) | 0.50 (0.577) | 0.54 (0.660) | 0.53 (0.624)

29. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response
Description: as for outcome 3
Time Frame: Week 2, 4, 8, 12, 20, 28, 40, 52
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Percentage of participants
  Week 2 | 0.0 | 62.5 | 41.7
  Week 4 | 50.0 | 75.0 | 66.7
  Week 8 | 75.0 | 100 | 91.7
  Week 12 | 100 | 87.5 | 91.7
  Week 20 | 100 | 87.5 | 91.7
  Week 28 | 100 | 100 | 100
  Week 40 | 75.0 | 100 | 91.7
  Week 52 | 50.0 | 100 | 83.3

30. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: greater than or equal to (>=) 50 percent (%) improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Percentage of participants
  Week 2 | 0.0 | 25.0 | 16.7
  Week 4 | 25.0 | 50.0 | 41.7
  Week 8 | 50.0 | 62.5 | 58.3
  Week 12 | 75.0 | 75.0 | 75.0
  Week 16 | 75.0 | 87.5 | 83.3
  Week 20 | 100 | 87.5 | 91.7
  Week 28 | 100 | 75.0 | 83.3
  Week 40 | 75.0 | 87.5 | 83.3
  Week 52 | 50.0 | 87.5 | 75.0

31. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: greater than or equal to (>=) 70 percent (%) improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Percentage of participants
  Week 2 | 0.0 | 0.0 | 0.0
  Week 4 | 0.0 | 37.5 | 25.0
  Week 8 | 25.0 | 62.5 | 50.0
  Week 12 | 50.0 | 62.5 | 58.3
  Week 16 | 50.0 | 62.5 | 58.3
  Week 20 | 75.0 | 75.0 | 75.0
  Week 28 | 75.0 | 50.0 | 58.3
  Week 40 | 50.0 | 75.0 | 66.7
  Week 52 | 50.0 | 75.0 | 66.7

32. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Component_ Tender/Painful Joint Count
Description: Sixty eight (68) joints were assessed by a rheumatologist investigator to determine the number of joints that were considered tender or painful. The response to pressure/motion on each joint was assessed with the following scale: Present/Absent/Not Done/Not Applicable (for Artificial or missing joints).
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: Psoriatic Arthritis Population: Participants who met the inclusion criteria for the psoriatic arthritis in the Full Analysis Set (FAS). FAS included all participants randomized and treated with at least 1 dose of study drugs.
Measure: Mean (Standard Deviation); unit: Tender/painful joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Tender/painful joints
  Week 2 | -1.8 (1.50) | -3.5 (2.78) | -2.9 (2.50)
  Week 4 | -6.3 (6.70) | -9.3 (11.37) | -8.3 (9.84)
  Week 8 | -11.5 (10.08) | -11.6 (10.24) | -11.6 (9.72)
  Week 12 | -13.8 (10.78) | -12.5 (11.95) | -12.9 (11.09)
  Week 16 | -13.0 (9.59) | -13.0 (12.17) | -13.0 (10.92)
  Week 20 | -14.3 (9.11) | -12.4 (12.87) | -13.0 (11.35)
  Week 28 | -14.0 (9.38) | -12.4 (12.52) | -12.9 (11.16)
  Week 40 | -14.3 (10.14) | -13.4 (12.09) | -13.7 (11.02)
  Week 52 (n=3, 8, 11) | -11.3 (9.24) | -13.5 (12.08) | -12.9 (10.97)

33. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Component_ Swollen Joint Count
Description: Sixty six (66) joints were assessed for swelling by a rheumatologist investigator to determine the number of joints that were considered swelling. The response to pressure/motion on each joint was assessed with the following scale: Present/Absent/Not Done/Not Applicable (for Artificial or missing joints).
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Swollen joints
  Week 2 | -1.8 (2.22) | -3.8 (5.55) | -3.1 (4.68)
  Week 4 | -5.0 (4.69) | -5.3 (5.80) | -5.2 (5.24)
  Week 8 | -6.0 (7.35) | -6.4 (4.37) | -6.3 (5.19)
  Week 12 | -6.5 (6.35) | -7.0 (4.44) | -6.8 (4.86)
  Week 16 | -7.3 (7.85) | -7.8 (3.85) | -7.6 (5.12)
  Week 20 | -7.0 (8.00) | -8.9 (4.42) | -8.3 (5.55)
  Week 28 | -7.3 (7.85) | -7.6 (4.03) | -7.5 (5.21)
  Week 40 | -7.3 (7.85) | -8.8 (4.20) | -8.3 (5.34)
  Week 52 (n=3, 8, 11) | -3.0 (0.00) | -8.8 (4.13) | -7.2 (4.38)

34. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Component_ Patient Assessment of Arthritis Pain
Description: Subjects assessed the severity of their arthritis pain with a 100 mm visual analog scale (VAS) by placing a mark on the scale between 0 (no pain) and 100 (the most severe pain), which corresponded to the magnitude of their pain.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Units on a scale
  Week 2 | -13.3 (8.30) | -29.5 (23.40) | -24.1 (20.77)
  Week 4 | -13.0 (23.41) | -41.4 (25.29) | -31.9 (27.42)
  Week 8 | -16.0 (19.78) | -43.6 (22.68) | -34.4 (24.88)
  Week 12 | -34.5 (19.71) | -46.0 (23.42) | -42.2 (22.07)
  Week 16 | -27.3 (15.22) | -46.0 (22.44) | -39.8 (21.65)
  Week 20 | -44.0 (22.82) | -45.3 (21.53) | -44.8 (20.91)
  Week 28 | -45.8 (23.26) | -45.8 (20.46) | -45.8 (20.34)
  Week 40 | -20.0 (54.86) | -46.9 (22.66) | -37.9 (36.37)
  Week 52 (n=3, 8, 11) | -33.0 (31.19) | -48.4 (22.14) | -44.2 (24.28)

35. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Component_ Patient Global Assessment of Arthritis
Description: Subjects answered the following question, "Considering the possible effects of the arthritis, how are you feeling today?" The subject's response was recorded with a 100 mm visual analog scale (VAS), where 0 = very well and 100 = very poorly.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Units on a scale
  Week 2 | -8.0 (8.87) | -32.6 (27.55) | -24.4 (25.53)
  Week 4 | -20.5 (11.27) | -43.4 (27.47) | -35.8 (25.33)
  Week 8 | -23.3 (19.69) | -51.3 (20.53) | -41.9 (23.75)
  Week 12 | -45.0 (8.83) | -52.1 (21.35) | -49.8 (17.99)
  Week 16 | -40.0 (13.64) | -53.0 (20.96) | -48.7 (19.27)
  Week 20 | -49.5 (20.09) | -49.6 (20.26) | -49.6 (19.27)
  Week 28 | -52.3 (11.18) | -46.3 (26.67) | -48.3 (22.26)
  Week 40 | -20.8 (30.24) | -50.8 (20.78) | -40.8 (27.24)
  Week 52 (n=3, 8, 11) | -40.7 (16.80) | -55.3 (20.51) | -51.3 (19.94)

36. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Component_ Physician Global Assessment of Arthritis
Description: The rheumatologist investigator assessed how the subject's overall arthritis appeared at the time of the visit. This was an evaluation based on the subject's disease signs, functional capacity and physical examination, and was independent of the PGA of arthritis. The rheumatologist investigator's response was recorded a 100 mm visual analog scale (VAS), where 0 = very good and 100 = very poor.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Units on a scale
  Week 2 | -15.3 (18.01) | -28.5 (18.60) | -24.1 (18.74)
  Week 4 | -32.5 (22.28) | -34.6 (19.39) | -33.9 (19.38)
  Week 8 | -29.5 (30.01) | -41.8 (21.87) | -37.7 (24.21)
  Week 12 | -39.8 (21.00) | -45.8 (22.76) | -43.8 (21.42)
  Week 16 | -49.8 (23.34) | -47.9 (20.09) | -48.5 (20.16)
  Week 20 | -50.8 (25.29) | -45.3 (26.81) | -47.1 (25.28)
  Week 28 | -49.5 (25.96) | -42.8 (22.79) | -45.0 (22.92)
  Week 40 | -38.5 (39.03) | -49.5 (18.54) | -45.8 (25.76)
  Week 52 (n=3, 8, 11) | -29.0 (20.30) | -46.8 (25.08) | -41.9 (24.32)

37. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Component_ C-Reactive Protein (CRP)
Description: The blood samples were collected at each visit for analysis of CRP with an assay analyzed by the central laboratory.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
mg/dL
  Week 2 | -1.20 (2.137) | -1.68 (2.231) | -1.52 (2.114)
  Week 4 | -1.20 (2.267) | -1.69 (2.272) | -1.53 (2.178)
  Week 8 | -1.28 (2.354) | -1.70 (2.222) | -1.56 (2.167)
  Week 12 | -1.28 (2.351) | -1.68 (2.235) | -1.54 (2.174)
  Week 16 | -1.30 (2.337) | -1.69 (2.189) | -1.56 (2.139)
  Week 20 | -1.33 (2.387) | -1.59 (2.336) | -1.50 (2.246)
  Week 28 | -1.30 (2.337) | -1.15 (2.770) | -1.20 (2.526)
  Week 40 (n=4, 7, 11) | -1.15 (2.037) | -1.84 (2.461) | -1.59 (2.236)
  Week 52 (n=3, 8, 11) | -0.03 (0.058) | -1.65 (2.295) | -1.21 (2.064)

38. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Component_ Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0=least difficulty and 3=extreme difficulty.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 40, 52
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Number analyzed (Participants) | 4 | 8 | 12
Units on a scale
  Week 2 | -0.19 (0.239) | -0.28 (0.376) | -0.25 (0.329)
  Week 4 | -0.28 (0.329) | -0.36 (0.381) | -0.33 (0.351)
  Week 8 | -0.28 (0.359) | -0.42 (0.433) | -0.38 (0.399)
  Week 12 | -0.28 (0.359) | -0.42 (0.433) | -0.38 (0.399)
  Week 16 | -0.31 (0.375) | -0.42 (0.433) | -0.39 (0.400)
  Week 20 | -0.28 (0.359) | -0.42 (0.433) | -0.38 (0.399)
  Week 28 | -0.34 (0.400) | -0.42 (0.433) | -0.40 (0.405)
  Week 40 | -0.09 (0.640) | -0.42 (0.433) | -0.31 (0.507)
  Week 52 (n=3, 8, 11) | -0.13 (0.573) | -0.42 (0.433) | -0.34 (0.465)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Total
Serious Adverse Events (participants affected / at risk) | 3/47 | 3/47 | 6/94
Other Adverse Events (participants affected / at risk) | 37/47 | 40/47 | 77/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=47) | CP-690,550 10 mg BID (N=47) | Total (N=94)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 3 | 0 | 3
Impetigo (Infections and infestations) | 0 | 1 | 1
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=47) | CP-690,550 10 mg BID (N=47) | Total (N=94)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 2
Asthenopia (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Conjunctival deposit (Eye disorders) | 0 | 1 | 1
Eyelid oedema (Eye disorders) | 1 | 0 | 1
Presbyopia (Eye disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Dental caries (Gastrointestinal disorders) | 3 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Lip erosion (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 2
Malaise (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 2 | 3
Pyrexia (General disorders) | 0 | 3 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 2 | 4
Bronchitis (Infections and infestations) | 1 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 2 | 2 | 4
Furuncle (Infections and infestations) | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 3 | 0 | 3
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 2
Herpes zoster (Infections and infestations) | 3 | 10 | 13
Hordeolum (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 3 | 3 | 6
Nasopharyngitis (Infections and infestations) | 14 | 14 | 28
Oral herpes (Infections and infestations) | 0 | 1 | 1
Otitis media acute (Infections and infestations) | 1 | 1 | 2
Periodontitis (Infections and infestations) | 0 | 1 | 1
Pertussis (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 1
Salpingitis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1
Tinea infection (Infections and infestations) | 1 | 1 | 2
Tinea pedis (Infections and infestations) | 4 | 6 | 10
Tinea versicolour (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Vaginitis gardnerella (Infections and infestations) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 5
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 3
Haemoglobin decreased (Investigations) | 1 | 4 | 5
Liver function test abnormal (Investigations) | 0 | 2 | 2
Low density lipoprotein increased (Investigations) | 0 | 1 | 1
Occult blood positive (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 3 | 3
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 2
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 4 | 6 | 10
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Solar dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Hypertension (Vascular disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.